## Statistical analysis

| Title of the study NTC Number | The Effect of GLP-1 Agonists Versus OCs on Reproductive Disorders and Cardiovascular Risks in Overweight PCOS NCT03151005 |
|---|---|
| Statistical method | Statistical analyses were performed using SPSS 23.0 and GraphPad Prism 8. For normally distributed con tinuous variables of clinical parameters, variables are described as the mean ± standard deviation (SD), a paired t-test was used to compare pretreatment and posttreatment values of continuous variables in each of the treatment groups, and between-group differences were compared by an independent sample t-te st. For nonnormally distributed continuous variables, the nonparametric Wilcoxon signed-rank test for rel ated samples was used to compare pretreatment and posttreatment values in each of the treatment groups. The chi-square test was used for counting data. To compare the changes in clinical parameters between different treatment groups, the nonparametric Mann-Whitney test was used. Proteomic data analysis was described by proteomic data acquisition and analysis. Protein levels are described as the mean±sta ndard error of the mean (SEM), and a paired ttest was used to compare plasma protein levels measured by ELISA. Pvalues <0.05 were considered statistically significant. |
| <b>Document Date</b> | July 28, 2017 |

Table 1-Baseline and posttreatment characteristics of cliniccal parameters after 12-week of treatment.

CPA/EE+Met(n=30)

GLP-1 RA+Met(n=30)

Characteristics Baseline Baseline Posttreatment Posttreatment **Pvalue Pvalue Biometric features** Weight(kg) BMI (kg/m²) Waist(cm) WHR SBP(mm/Hg) DBP(mm/Hg **Reproductive function** Dominant follicle,n(%) Regular menstruation, n(%) Amenorrhoea, n(%)\* Oligomenorrhoea,n(%)+ Polycystic ovaries according t o Rotterdam criteria, n(%) T(nmol/L) LH(mlU/ml) FSH(mIU/mI) LH/FSH DHEA-S(ug/dL) SHBG (nmol/L) FAI E2(pg/ml) P(ng/ml) PRL(ng/ml) Biochemical profile of glucose metabolism HbA1c(%) HbA1c(mmol/mol) FBG(mmol/L) **AUCI** FINS(uU/ml) **HOMA-IR** Biochemical profile of lipid metabolism TG(mmol/L)

Data are mean±SD orn(%). BMI, body mass index; WHR, waist-to-hip ratio; SBP, systolic blood pressure; DBP, diastolic blood pressure; T, testerone; LH, luteinizing hormone; FSH, follicle- stimulating hormone; DHEA-S, dehydroepiandrosterone; SHBG, sex hormone-binding globulin; FAI, free androgen index; E2, estradiol; P, progesterone; PRL, prolactin. HbA1c, hemoglobin A1c; FBG, fasting blood gl ucose; FINS, fasting insulin; AUCI, area under curve of insulin; HOMA- IR, homoeostasis model assessment of insulin resistance; T G, triglycerides; TC, total cholesterol

TC(mmol/L)

GLP-1 RA +Met

(n=30)

t/z

Pvalue

CPA/EE +Met Characteristics (n=30)Biometric features  $\triangle$ Weight(kg)  $\triangle$ BMI (kg/m $^2$ ) △Waist(cm)  $\triangle$ WHR  $\triangle$ SBP (mm/Hg)  $\triangle$ DBP (mm/Hg) Sex hormones and related indicators  $\triangle T (nmo1/L)$  $\triangle$ LH(m1U/m1) AFSH (m1U/m1) ALH/FSH  $\triangle$ DHEA-S (ug/dL) △SHBG (nmo1/L)△FAI  $\triangle$ E2(pg/m1)  $\triangle P(ng/m1)$  $\triangle$ PRL (ng/m1)  $Biochemical\ profile\ of\ lipid\ metabolism$ 

 $\triangle$ TG (mmo1/L)

 $\triangle$ TC (mmo1/L)